CLINICAL TRIAL: NCT04406740
Title: Clinical Evaluation of a Novel Neuromuscular Blockade Monitoring System
Status: Terminated | Type: Observational
Why Stopped: Device malfunction
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: ANES-2020-28905
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Participants: Adult patients >18 years of age, who are scheduled to undergo any elective procedure under general anesthesia in the MHealth East Bank operating rooms in which the administration of a nondepolarizing neuromuscular blocking drug (rocuronium or cisatracurium) is anticipated.
  Interventions: Device: TwitchView EMG Unit; Device: Novel QTOF Device

INTERVENTIONS:
Device: TwitchView EMG Unit — The TwitchView device is a new generation electromyographic monitor that uses a disposable electrode array that combines stimulating and recording electrodes.
Device: Novel QTOF Device — The QTOF consists of an electrical stimulator that is just like the stimulator in the traditional TOF devices that are commonly used (both accelerometric and EMG-based), combined with a novel sensor that sticks to the belly of the muscle being measured (most commonly the adductor pollicis, the thumb muscle in the palm of the hand).

SUMMARY:
This study is designed to formally evaluate the performance of the QTOF, as compared with the newest commercially available NMB monitoring equipment, EMG (the TwitchView).

DETAILED DESCRIPTION:
The disposable stimulus/recording electrode array for the TwitchView will be placed on one of the patient's wrist/hand and connected to the device. Next, the stimulating electrodes and vibration sensor of the QTOF device will be placed over the contralateral ulnar nerve and thenar eminence. The devices will be placed prior to the induction of anesthesia - but no electrical stimuli will be delivered until AFTER the patient is asleep (as per routine). After induction, both devices will be started. The TwitchView automatically selects the appropriate stimulus current (takes about 10 seconds) - and when that is complete, the QTOF stimulus current will be set to the same value. The stimulus interval for both devices will be 20 seconds. Paired measurements of twitch count and TOF ratios will be gathered for the entirety of the surgical procedure, and cross checked with Epic regarding the administration of neuromuscular blocking drugs (time, dose) and reversal agents (time, dose). RAs will be present to verify the correct function of both devices. Note that information from the TwitchView monitor will be continuous available to the providers (it is a standard device available for use in our ORs). Information from the QTOF will NOT be made available to providers.

ELIGIBILITY:
Inclusion Criteria:

- patients scheduled to undergo any elective procedure under general anesthesia in the MHealth East Bank operating rooms in which the administration of a nondepolarizing neuromuscular blocking drug (rocuronium or cisatracurium) is anticipated

Exclusion Criteria:

* Emergent procedures will be excluded
* Procedures performed outside of regular Monday to Friday working hours will be excluded
* Inability to provide their own consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients >18 years of age, who are scheduled to undergo any elective procedure under general anesthesia in the MHealth East Bank operating rooms in which the administration of a nondepolarizing neuromuscular blocking drug (rocuronium or cisatracurium) is anticipated.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Train-of-Four (TOF) Ratio | 420 minutes
  The train-of-four ratio (unitless measure) is calculated by comparing the magnitude of the fourth evoked response or twitch (T4) to that of the first response (T1).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Todd, MD, Principal Investigator — University of Minnesota
Locations (1):
- MHealth Farview University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided